CLINICAL TRIAL: NCT04047914
Title: Antimicrobial Photodynamic Therapy in the Nasal Decolonization of Maintenance Hemodialysis Patients: A Pilot Randomized Trial
Brief Title: Antimicrobial Photodynamic Therapy in the Nasal Decolonization of Maintenance Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Anna Carolina Ratto Tempestini Horliana, Phd, clinical professor, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NASAL DECOLONIZATION
Record Dates: First submitted 2019-08-02; First posted 2019-08-07 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-01

CONDITIONS: Photochemotherapy; Renal Insufficiency, Chronic
Keywords: antimicrobial photodynamic therapy; Staphylococcus aureus; nasal decolonization; hemodialysis; chronic kidney disease; mupirocin
MeSH Terms: conditions — Renal Insufficiency, Chronic; Staphylococcal Infections | interventions — Photochemotherapy

STUDY DESIGN:
Intervention Model Description: 34 individuals will be randomly divided into 2 groups: G1 - Experimental Group (n = 17) - Treatment will be performed with methylene blue and red light-emitting diode (LED) in the nostrils. G2 - Control group (n = 17) - Standard treatment will be performed conventionally with topical mupirocin.
Who Masked: Outcomes Assessor
Masking Description: The researcher responsible for performing the treatments (which will open the randomization envelopes) will know which treatment is assigned to each patient. The researcher responsible for collecting the microbiological samples (nasal discharge) and the microbiologist will be blind to the treatments assigned to the groups (they do not know the nature of treatments). The patient will not be blinded in view of the difference between the nature of the treatments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental aPDT group (Experimental): Application of 0.01% methylene blue with enough sterile swab to cover the inner nostril extension with a 10 minute pre-irradiation time. The irradiations were carried out with a red light-emitting diode (LED) (λ = 660 nm), for 300 seconds, irradiance of 400 mW / cm2, radiant exposure 124 J / cm2, with uniform application in each anterior nostril.
  Interventions: Device: Antimicrobial Photodynamic therapy
- control mupirocin group (Active Comparator): A standard treatment will be performed conventionally with topical mupirocin. Will be performed with 2% Mupirocin Ointment, to be applied to the anterior nostrils twice a day for 5 days.
  Interventions: Drug: Mupirocin ointment

INTERVENTIONS:
Device: Antimicrobial Photodynamic therapy — Application 0.01% methylene blue with sterile swabs in each nostril with a 10-minute pre-irradiation
  • Light-emitting diode (λ = 660 nm), for 300 seconds, with an irradiance of 400 mW / cm2
  Other Names: Photochemotherapy
  Arms: experimental aPDT group
Drug: Mupirocin ointment — Performed with 2% Mupirocin Ointment, to be applied to the anterior nostrils twice a day for 5 days.
  Other Names: Mupirocin Nasal Product
  Arms: control mupirocin group

SUMMARY:
The objective of this study will be to evaluate the effect of Antimicrobial Photodynamic Therapy (aPDT) in the Nasal Decolonization of Dialytic Chronic Renal Patients, Staphylococcus Aureus (S.aureus) Carriers This is a 3-months follow-up, randomized, single-blind, prospective controlled trial, single-center and will happen in 02 phases: Phase 1 - Epidemiological Evaluation - A researcher will invite the research participants who are undergoing treatment at the Hemodialysis Service of Clinical Hospital and explain its contents. After reading and signing the informed consent, this same researcher (calibrated for the experiment) will perform nasal secretion microbiological collections to identify patients colonized by S.aureus in the anterior nostril (nasal carrier) - baseline T0 and the application of the questionnaire that identifies possible factors that may be considered as risk for colonization and possible development of diseases related to S. aureus. In the laboratory of Microbiology, the strains will be identified and the colonized patients will be invited to continue the study (Phase 2). Non-carrier patients will only be counseled with infection prevention care. Phase 2 - Parallel clinical trial with two intervention groups (aPDT or Mupirocin) - Patients with nasal aureus (thirty-four colonized patients aged over 18 years) will be treated with aPDT (experimental group) or mupirocin (control group). A trained researcher will collect new aliquots of nasal discharge after completion of nostril treatment (T1) to check for decolonization by culture. A new collection will be performed at 1 (T2) and 3 (T3) months after treatment to assess recolonization. It was evaluated intervention safety (photodynamic therapy) through a directed and open questionnaire about adverse effects.

DETAILED DESCRIPTION:
Infections are the leading cause of morbidity and the second leading cause of mortality among patients with chronic kidney disease (CKD) on renal replacement therapy. Staphylococcus aureus (S. aureus) is a major agent and previous nasal colonization represents an independent risk factor for infection. Up to 50% of these patients can be known to be colonized. With the global increase in bacterial resistance by S.aureus strategies for infection prevention and transmission by this agent are needed. The strategy of decolonization and elimination of nasal carrier status by S.aureus in dialytic chronic renal patients reduces infection rates, especially bacteremia. The gold standard for nasal decolonization is topical mupirocin treatment, but there are reports of increasing resistance especially after prolonged use, which limits the establishment of clinical protocols for the prevention of infection in the dialysis population. Antimicrobial Photodynamic Therapy (aPDT) proves to be a promising approach for its potential bactericidal effect, including multidrug-resistant bacteria and its low tendency to induce drug resistance.

This is a 3-months follow-up, randomized, single-blind, prospective controlled trial, single-center and will happen in 02 phases: Phase 1 - Epidemiological Evaluation - A researcher will invite the research participants who are undergoing treatment at the Hemodialysis Service of Clinical Hospital and explain its contents. After reading and signing the informed consent, this same researcher (calibrated for the experiment) will perform nasal secretion microbiological collections to identify patients colonized by S.aureus in the anterior nostril (nasal carrier) - baseline T0 and the application of the questionnaire that identifies possible factors that may be considered as risk for colonization and possible development of diseases related to S. aureus. In the laboratory of Microbiology, the strains will be identified and the colonized patients will be invited to continue the study (Phase 2). Non-carrier patients will only be counseled with infection prevention care. Phase 2 - Parallel clinical trial with two intervention groups (aPDT or Mupirocin) - Patients with nasal aureus (thirty-four colonized patients aged over 18 years) will be treated with aPDT (experimental group) or mupirocin (control group). Two other trained researchers will collect new aliquots of nasal discharge after completion of nostril treatment (T1) to check for decolonization by culture. A new collection will be performed at 1 (T2) and 3 (T3) months after treatment to assess recolonization.It was evaluated intervention safety (photodynamic therapy) through a directed and open questionnaire about adverse effects,immediately after treatments, with a 3-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* nasal carriers of S.aureus
* chronic kidney patient undergoing hemodialysis treatment;
* aged over 18 years;
* both genders;

Exclusion Criteria:

* pregnancy or breastfeeding;
* presence of nasal foreign body;
* history of nasal surgery in the last 3 months;
* active infection by S. aureus;
* use of topical nasal or systemic antibiotic in the last three months;
* history of severe allergy to mupirocin or methylene blue (MB);

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-07-12 (Actual)

PRIMARY OUTCOMES:
Qualitative culture (presence or absence bacterial colonies) after aPDT (antimicrobial photodynamic therapy) decolonization or mupirocin | Before the intervention (T0)
  The microbiological analysis was done by MALDI-TOF (Biomérieux) - Matrix Associated Laser Desorption-Ionization - Time of Fligh
Qualitative culture (presence or absence bacterial colonies) after aPDT (antimicrobial photodynamic therapy) decolonization or mupirocin | Immediately after the completion of treatments (T1)
  The microbiological analysis was done by MALDI-TOF (Biomérieux) - Matrix Associated Laser Desorption-Ionization - Time of Fligh

SECONDARY OUTCOMES:
Prevalence of S.aureus | initial screening time to assess nasal staphylococcus aureus carrier before treatments
  To evaluate the prevalence of both sensitive and methicillin-resistant S.aureus patients by bacterial culture and antibiogram in patients with renal chronic disease on dialysis treatment at the Hemodialysis Service of the University of São Paulo Medical School of Sao Paulo.
Prevalence of recolonization | 01 and 03 months after treatments
  To evaluate the prevalence of recolonization by Staphylococcus aureus in the anterior nostril in through qualitative microbiological culture (presence or absence). The microbiological analysis was done by MALDI-TOF (Biomérieux) - Matrix Associated Laser Desorption-Ionization - Time of Flight.
Anamnesis and risk factor collection | immediately after recruiting and accepting patients who met the inclusion/exclusion criteria
  Guiding questions were applied to all patients. In addition to questions related to the patient's general health, demographic data (age, gender, marital status, occupation, education, housing), medical history data (etiology of CKD ( renal chronic disease), comorbidities, time of dialysis treatment until protocol initiation, presence smoking rate, type of venous access and time of use, kidney transplantation, systemic antibiotic therapy in the last 12 months, hospitalization or infection (including skin) in the last 12 months).
Ontervention safety: photodynamic therapy | immediately after treatments, with a 3-month follow-up
  The analysis of adverse effects through a directed and open questionnaire, especially for this study

CONTACTS AND LOCATIONS:
Overall Officials: Anna Carolina RT Horliana, phD, Principal Investigator — Nove de Julho University; Daniella T Bezerra, phD, Principal Investigator — Nove de Julho University
Locations (1):
- University of Nove de Julho (UNINOVE), São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fu XJ, Fang Y, Yao M. Antimicrobial photodynamic therapy for methicillin-resistant Staphylococcus aureus infection. Biomed Res Int. 2013;2013:159157. doi: 10.1155/2013/159157. Epub 2013 Feb 28. PMID 23555074
- [Result] Wertheim HF, Melles DC, Vos MC, van Leeuwen W, van Belkum A, Verbrugh HA, Nouwen JL. The role of nasal carriage in Staphylococcus aureus infections. Lancet Infect Dis. 2005 Dec;5(12):751-62. doi: 10.1016/S1473-3099(05)70295-4. PMID 16310147
- [Result] Tacconelli E, Carmeli Y, Aizer A, Ferreira G, Foreman MG, D'Agata EM. Mupirocin prophylaxis to prevent Staphylococcus aureus infection in patients undergoing dialysis: a meta-analysis. Clin Infect Dis. 2003 Dec 15;37(12):1629-38. doi: 10.1086/379715. Epub 2003 Nov 20. PMID 14689344
- [Derived] Bezerra DT, La Selva A, Cecatto RB, Deana AM, Prates RA, Bussadori SK, Mesquita-Ferrari RA, Motta LJ, Fernandes KPS, Martimbianco ALC, Frochot C, Pereira BJ, Rossi F, Mimica MJ, Horliana ACRT. Antimicrobial Photodynamic Therapy in the Nasal Decolonization of Maintenance Hemodialysis Patients: A Pilot Randomized Trial. Am J Kidney Dis. 2023 May;81(5):528-536.e1. doi: 10.1053/j.ajkd.2022.09.013. Epub 2022 Nov 14. PMID 36396084